CLINICAL TRIAL: NCT04925739
Title: Evaluation of the Comfort of a Continuous Positive Airway Pressure Nasal Mask in the Treatment of Obstructive Sleep Apnea Syndrome
Brief Title: Evaluation of the Comfort of a Continuous Positive Airway Pressure Nasal Mask in the Treatment of OSA Syndrome
Acronym: NINADOM
Status: Completed | Type: Observational
Sponsor: AGIR à Dom (Other)
Collaborators: Air Liquide SA (Industry)
Responsible Party: Sponsor
Other Study IDs: RCB : 2021-A01510-41
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-01

CONDITIONS: Apnea, Obstructive
Keywords: Obstructive Sleep Apnea; Continuous Positive Airway Pressure; Mask
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OSA patients treated with CPAP: OSA patient, not previously treated with CPAP, are treated with a "ResMed Airsense 10" CPAP and an "Air Liquide Medical Systems" NINA mask during 30 days, monitored by the home care provider AGIRADOM.
  After 30 days of CPAP treatment, 4 self-questionnaires are completed by the patient and parameters of the CPAP treatment (compliance, estimated unintentional leakage and therapeutic pressures) are collected.
  Interventions: Other: Self-questionnaire on the comfort and general appreciation of a nasal mask; Other: Self-questionnaire on the appearance of CPAP side effects related to the mask; Other: Self-questionnaire on the patient's appreciation of the mask headgear,; Other: Self-questionnaire NOSE on the discomfort caused by the nasal obstruction; Other: Self-questionnaire Epworth on the daytime sleepiness; Other: To study the CPAP compliance; Other: To study the unintentional leakage; Other: To study the therapeutic pressures of CPAP

INTERVENTIONS:
Other: Self-questionnaire on the comfort and general appreciation of a nasal mask — Self-questionnaire on the comfort and general appreciation of a nasal mask after 30 days of use
Other: Self-questionnaire on the appearance of CPAP side effects related to the mask — Self-questionnaire on the appearance of CPAP side effects related to the mask (air leaks, injury to the nasal bridge, etc.) after 30 days of use
Other: Self-questionnaire on the patient's appreciation of the mask headgear, — Self-questionnaire NOSE (Nasal Obstruction Symptom Evaluation) on the patient's appreciation of the mask headgear, which includes indications to help with the installation in the form of graduated markers, as well as the appreciation of the general aesthetics of the mask, after 30 days of use.
Other: Self-questionnaire NOSE on the discomfort caused by the nasal obstruction — Self-questionnaire NOSE on the discomfort caused by the nasal obstruction reported by the patient, after 30 days of use, compared to the inclusion.
Other: Self-questionnaire Epworth on the daytime sleepiness — Self-questionnaire Epworth on the daytime sleepiness of the patient, after 30 days of treatment, compared to the inclusion.
  To study the parameters of the CPAP treatment.
Other: To study the CPAP compliance — To collect the treatment compliance through telemonitoring of the data recorded by the CPAP machine, during the 30 days of treatment.
Other: To study the unintentional leakage — To collect the unintentional leakage estimated by the CPAP machine, during the 30 days of treatment.
Other: To study the therapeutic pressures of CPAP — To collect the therapeutic pressures of CPAP, during the 30 days of treatment.

SUMMARY:
Continuous positive airway pressure (CPAP) is the first-line treatment for obstructive sleep apnea syndrome (OSA). It consists of a pressure generator connected to a mask applied to the patient's face. CPAP treatment is restrictive, and nearly a quarter of patients abandon it over the long term. Various factors can influence adherence to CPAP therapy, including adverse events associated with the mask. However, it is clear that compliance with CPAP treatment, even if it has tended to improve over the last 30 years, is still sub-optimal.

The "Air Liquide Medical Systems" company has developed a mask that aims to improve comfort and ease of use for the patient. This leaky nasal mask has a "silent" intentional leak port, which significantly reduces the noise caused by the escape of air. The noise associated with intentional leakage is one of the discomforts reported by patients and their spouses. In addition, this mask is equipped with a new generation headgear with adjustment indicators to assist the patient in fitting the mask. Optimal headgear fit is a prerequisite for comfort during treatment, as it reduces unintentional leakage.

The main objective is to evaluate, through a questionnaire, the comfort and general appreciation of a nasal mask equipped with a silent leak system and a headgear with adjustment aids, of patients with OSA treated with CPAP.

Secondary objectives are :

1. To evaluate the appearance of CPAP side effects related to the mask,
2. To collect the patient's appreciation of the mask headgear,
3. To evaluate the discomfort caused by the nasal obstruction reported by the patient,
4. To evaluate the daytime sleepiness of the patient,
5. To study the parameters of the CPAP treatment.

DETAILED DESCRIPTION:
Continuous positive airway pressure (CPAP) is the first-line treatment for obstructive sleep apnea syndrome (OSA). It consists of a pressure generator connected to a mask applied to the patient's face. CPAP treatment is restrictive, and nearly a quarter of patients abandon it over the long term. Various factors can influence adherence to CPAP therapy, including adverse events associated with the mask. Unintentional leaks, i.e. a leak between the pressure generator and the patient's upper airway, are among the most frequent. Therefore, optimizing the choice of mask is one of the main means used by medical-technical providers, in charge of installing CPAP and its technical follow-up at home. In order to cover the needs and anatomical particularities of the OSA patient population treated with CPAP, a large number of mask types and sizes are currently available on the market. However, it is clear that compliance with CPAP treatment, even if it has tended to improve over the last 30 years, is still sub-optimal.

The "Air Liquide Medical Systems" company has developed a mask that aims to improve comfort and ease of use for the patient. This leaky nasal mask has a "silent" intentional leak port, which significantly reduces the noise caused by the escape of air. The noise associated with intentional leakage is one of the discomforts reported by patients and their spouses. In addition, this mask is equipped with a new generation headgear with adjustment indicators to assist the patient in fitting the mask. Optimal headgear fit is a prerequisite for comfort during treatment, as it reduces unintentional leakage.

The main objective is to evaluate, through a questionnaire, the comfort and general appreciation of a nasal mask equipped with a silent leak system and a headgear with adjustment aids, of patients with OSA treated with CPAP.

After 30 days of use, secondary objectives are :

1. To evaluate the appearance of CPAP side effects related to the mask (air leaks, injury to the nasal bridge, etc.)
2. To collect the patient's appreciation of the mask headgear, which includes indications to help with the installation in the form of graduated markers, as well as the appreciation of the general aesthetics of the mask.
3. To evaluate the discomfort caused by the nasal obstruction reported by the patient, in relation to the inclusion.
4. To evaluate the daytime sleepiness of the patient, compared to the inclusion.
5. To study the parameters of the CPAP treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient over 18 years of age
* Patient with OSA
* Patient not previously treated with CPAP
* A patient who will be treated with a "ResMed Airsense 10" CPAP and an "Air Liquide Medical Systems" NINA mask
* Patient whose CPAP treatment will be installed and monitored by the home care provider AGIRADOM
* Patient willing to participate in the research after adequate information and delivery of the information note
* Patient affiliated to the social security system or beneficiary of such a system

Exclusion Criteria:

* NOSE questionnaire score greater than or equal to 10/20 at the time of CPAP installation
* Patient with significant craniofacial deformities that do not allow the mask to be fitted correctly
* Person deprived of liberty by judicial or administrative decision, person under legal protection (patient under guardianship or curators) Article L1121-8
* Subject who receives more than 4500 euros in compensation for his or her participation in other research involving the human person in the 12 months preceding this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: OSA patient, not previously treated with CPAP, who will be treated with a ResMed Airsense 10 CPAP and an Air Liquide Medical Systems NINA mask Patient whose CPAP treatment will be installed and monitored by the home care provider AGIRADOM.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
To evaluate the comfort and general appreciation of a nasal mask | After 30 days of CPAP treatment
  to evaluate, through a questionnaire, the comfort and general appreciation of a nasal mask equipped with a silent leak system and a headgear with adjustment aids, of patients with OSA treated with CPAP.

SECONDARY OUTCOMES:
To evaluate the appearance of CPAP side effects related to the mask | After 30 days of CPAP treatment
  To evaluate the appearance of CPAP side effects, through a questionnaire, related to the mask (air leaks, injury to the nasal bridge, etc.)
To collect the patient's appreciation of the mask headgear | After 30 days of CPAP treatment
  To collect, through a questionnaire, the patient's appreciation of the mask headgear, which includes indications to help with the installation in the form of graduated markers, as well as the appreciation of the general aesthetics of the mask.
To evaluate the discomfort caused by the nasal obstruction reported by the patient | After 30 days of CPAP treatment
  To evaluate, trough the NOSE questionnaire, the discomfort caused by the nasal obstruction reported by the patient, compared to the inclusion.
To evaluate the daytime sleepiness of the patient | After 30 days of CPAP treatment
  To evaluate the daytime sleepiness of the patient, through the Epworth questionnaire, compared to the inclusion.
To collect the CPAP treatment compliance | During the 30 days of CPAP treatment
  To collect the treatment compliance (average daily use) through telemonitoring of the data recorded by the CPAP machine.
To collect the unintentional leakage | During the 30 days of CPAP treatment
  To collect the unintentional leakage estimated by the CPAP machine.
To collect the CPAP therapeutic pressures | During the 30 days of CPAP treatment
  To collect the CPAP therapeutic pressures used.

CONTACTS AND LOCATIONS:
Overall Officials: LEBRET Marius, Study Director — AIR LIQUIDE MEDICAL SYSTEMS
Locations (1):
- Pauline Socquet, Meylan, France